CLINICAL TRIAL: NCT06867926
Title: The Effect of Cardiac Rehabilitation on Oxidative DNA Damage and Inflammation in Patients With Coronary Artery Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Hasan Kara, Professor Assistant Medical Doctor, TC Erciyes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKara3
Record Dates: First submitted 2024-10-16; First posted 2025-03-10 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: Cardiac Rehabilitation; Oxidative DNA damage; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group for cardiac rehabilitation with coronary artery disease (Experimental): Individuals diagnosed with coronary artery disease will engage in a programme of cardiac rehabilitation.
  Interventions: Other: Cardiac rehabilitation
- Healthy control group (No Intervention)

INTERVENTIONS:
Other: Cardiac rehabilitation — Individuals diagnosed with coronary artery disease will engage in a programme of cardiac rehabilitation.
  Arms: Study group for cardiac rehabilitation with coronary artery disease

SUMMARY:
The objective of this study was to determine the levels of 8-hydroxy-2'-deoxyguanosine (8-OHdG), an indicator of oxidative stress, and to demonstrate oxidative DNA damage in cardiac rehabilitation treatment in patients with coronary artery disease. Additionally, proinflammatory cytokines TNFα, IL-1β, and IL-6 levels were measured to evaluate the significance of cardiac rehabilitation treatment in patients with coronary artery disease and to assess the correlation between cytokine levels and 8-OHdG levels.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is a significant global health issue and the leading cause of cardiovascular mortality.

Recent research has focused on the impact of oxidative stress, genetic damage, and inflammation in CAD development. Chronic inflammation and oxidative stress can cause cellular damage by increasing the formation of free oxygen radicals. Oxidative stress leads to endothelial dysfunction, inflammation of the vessel wall, and the formation of atherosclerotic plaques. Atherosclerosis is the most common pathological process associated with cardiovascular diseases, and the disease is characterized by a high oxidative stress state, which causes lipid and protein oxidation. Oxidative stress and an imbalance between oxidants and antioxidants can damage important biomolecules such as DNA, lipids, and proteins.

Cardiac rehabilitation (CR) programmes are a recommended therapy with demonstrated efficacy in the treatment of patients with CAD. CR is a holistic approach that combines medical and exercise interventions to improve patients' cardiovascular health and general well-being. Exercise is the foundation of CR. While the literature describes it extensively, there is still some controversy surrounding oxidative stress and exercise. It has been suggested that exercise may increase the production of reactive oxygen molecules associated with oxidative stress, which is a factor in the pathogenesis of CAD. Regular and moderate exercise can have a positive impact on the body by balancing the production of antioxidants, reducing inflammation and oxidative stress. However, it is important to note that exercise should be approached in moderation to avoid any negative effects on the body. Previous studies have focused on risk factors associated with physical fitness, the fibrinolytic system, or lipid profile in cardiac patients. However, there have been relatively few investigations of induced changes in blood.

This study aims to investigate the role of oxidative stress and inflammation in the pathogenesis of CAD and the effects of KR on these pathophysiological processes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Patient Volunteers

1. Patients aged 18-65 years with a diagnosis of coronary artery disease and no contraindications to cardiac rehabilitation and exercise testing
2. Patients who will undergo cardiopulmonary exercise testing before cardiac rehabilitation
3. Patients whose cognitive status is sufficient to complete the study and who can cooperate

Inclusion Criteria for Healthy Volunteers

1. 18 years of age or older
2. Not having a chronic disease (such as uncontrolled diabetes mellitus, hypertension, heart and kidney failure)
3. Not taking regular medication

Exclusion Criteria:

Exclusion Criteria for Patient Volunteers

1. Having heart failure
2. Unstable Angina Pectoris
3. Complex ventricular arrhythmia
4. Having a pacemaker
5. Having orthopedic or neurological diseases that prevent exercise
6. Having kidney-liver disease
7. Exercise is contraindicated
8. History of inflammatory diseases
9. Having a history of cancer-immunologic disease

Exclusion Criteria for Healthy Volunteers

1. Having a history of chronic diseases such as diabetes mellitus, hypertension, heart and kidney failure
2. Being on regular medication for the last 6 months
3. being under 18 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
8-OHdG | intervention group, two measurements- before cardiac rehabilitation (one day before the intervention) and two measurements will be taken after cardiac rehabilitation (at the end of the program)A single measurement will be performed on the healthy control
  To measure 8-OHdG in serum samples, the investigators will analyze it using the ELISA kit following the kit procedure and measure it on an ELISA reader.
NADPH oxidase (NOX) | intervention group, two measurements- before cardiac rehabilitation (one day before the intervention) and two measurements will be taken after cardiac rehabilitation (at the end of the program)A single measurement will be performed on the healthy control
  To measure NOX in serum samples, the investigators will analyze it using the ELISA kit following the kit procedure and measure it on an ELISA reader.
Total antioxidant capacity (TAC) | intervention group, two measurements- before cardiac rehabilitation (one day before the intervention) and two measurements will be taken after cardiac rehabilitation (at the end of the program)A single measurement will be performed on the healthy control
  To measure TAC in serum samples, the investigators will analyze it using the ELISA kit following the kit procedure and measure it on an ELISA reader.
Total oxidant status (TOS) | intervention group, two measurements- before cardiac rehabilitation (one day before the intervention) and two measurements will be taken after cardiac rehabilitation (at the end of the program)A single measurement will be performed on the healthy control
  To measure TOS in serum samples, the investigators will analyze it using the ELISA kit following the kit procedure and measure it on an ELISA reader.
Proinflammatory cytokines (TNFα, IL-1β and IL-6) | intervention group, two measurements- before cardiac rehabilitation (one day before the intervention) and two measurements will be taken after cardiac rehabilitation (at the end of the program)A single measurement will be performed on the healthy control
  To measure TNFα, IL-1β and IL-6 in serum samples, the investigators will analyze it using the ELISA kit following the kit procedure and measure it on an ELISA reader.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Medicine, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No